CLINICAL TRIAL: NCT04491695
Title: Safety and Efficacy of Tirofiban in Preventing Neurological Deterioration of Patients With Acute Ischemic Stroke: A Randomized Controlled Trial
Brief Title: Tirofiban for the Prevention of Neurological Deterioration in Acute Ischemic Stroke
Acronym: TREND
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Ji Xunming,MD,PhD, Professor, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TREND
Record Dates: First submitted 2020-07-25; First posted 2020-07-29 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Acute Stroke
Keywords: Acute ischemic stroke; Neurological deterioration; Stroke progression
MeSH Terms: conditions — Stroke; Ischemic Stroke | interventions — Tirofiban

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tirofiban+Oral antiplatelet therapy (Experimental): Patients will receive Tirofiban in the first 72 hours and bridge to oral antiplatelet therapy thereafter.
  Interventions: Drug: Tirofiban Hydrochloride; Drug: Oral antiplatelet
- Oral antiplatelet therapy (Active Comparator): Patients will receive oral antiplatelet therapy alone.
  Interventions: Drug: Oral antiplatelet

INTERVENTIONS:
Drug: Tirofiban Hydrochloride — Tirofiban will use a loading dose, 0.4 μg/kg/min × 30 minutes, then 0.1μg/kg/min infusion for 71.5 hours.
  Arms: Tirofiban+Oral antiplatelet therapy
Drug: Oral antiplatelet — Aspirin, clopidogrel or other antiplatelet drugs. Loading dose will be considered if the patients is not on antiplatelet therapy.

SUMMARY:
Currently, dual antiplatelet therapy with aspirin and clopidogrel (with loading doses) is widely used for patients with acute ischemic stroke. However, immediate, potent and reversible inhibition of platelet aggregation is not possible. Additionally, more than 5% patients have aspirin resistance and more than 15% patients have clopidogrel resistance. Therefore, an intravenously administered GPIIb/IIIa receptor inhibitor (Tirofiban) receptor blocker with fast onset and offset of actions will provide more desired antiplatelet effects in the setting of acute ischemic stroke, especially in patients with high risk of neurological deterioration. This study will measure the anti-platelet effects of Tirofiban in patients with acute ischemic stroke who had high risk of neurological deterioration.

ELIGIBILITY:
Inclusion Criteria:

1. Acute ischemic stroke with 24 hours of symptom onset.
2. NIHSS≥4 and ≤20 points, and the paralyzed limbs is able to actively move the muscle (standardized motor examination rating scale of 2 or much higher).
3. Age 18-80 years old.
4. Informed consent obtained from patient or acceptable patient's surrogate.

Exclusion Criteria:

1. Treated with intravenous or endovascular thrombectomy for the indexed acute ischemic stroke.
2. Acute ischemic stroke caused by determined or suspected cardioembolism.
3. Acute ischemic stroke caused by other determined caused, including moyamoya disease, artery dissection, arteritis, and etc.
4. Pre-stroke mRS ≥2 or the paralyzed limbs are dyskinesia before stroke.
5. Known hematochezia, gastrointestinal bleeding and any other bleeding.
6. Allergy to tirofiban or its solvents.
7. Patients suffered from severe diseases, including malignant tumor, liver cirrhosis, kidney failure, congestive heart failure, and etc.
8. Gastrointestinal or genitourinary tract bleeding within 1 years.
9. Determined coagulation disorders, platelet dysfunction, or platelet count <100*109/L.
10. Major surgical operation or severe trauma within 1 month.
11. Hemorrhagic retinopathy.
12. Chronic hemodialysis.
13. Uncontrolled hypertension with systolic blood pressure >180 mmHg or diastolic blood pressure >110 mmHg.
14. Acute pericarditis.
15. Other conditions that determined by the investigators.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2020-09-12 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients with a change in NIHSS by ≥ 4 points compared to enrollment NIHSS. | Within 72 hours of intervention.
  National Health Institute Stroke Scale (NIHSS): stroke symptom severity scale with a range of 0-42. Higher score means more severe stroke symptoms.

SECONDARY OUTCOMES:
Change of the NIHSS | 0-30 days of intervention.
  National Health Institute Stroke Scale (NIHSS): stroke symptom severity scale with a range of 0-42. Higher score means more severe stroke symptoms.
Change of the Scandinavian Stroke Scale | 0-30 days of intervention.
  Scandinavian Stroke Scale (SSS): stroke symptom severity scale with a range of 0-58. Lower score means more severe stroke symptoms.
The severity of global disability at 90 days, as assessed by modified Rankin scale (mRS). | 0-90 days.
  The mRS is an ordinal, graded interval scale that assigns patients among 7 global disability levels, which ranging from 0 (no symptom) to 5 (severe disability) and 6 (death).
Rate of symptomatic intracerebral hemorrhage. | 0-90 days
Number of Participants experienced adverse events | 0-90 days.

CONTACTS AND LOCATIONS:
Locations (19):
- China (19):
  - Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Luhe Hospital, Capital Medical University, Beijing, Beijing Municipality
  - The first Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - Nanyang Central Hospital, Nanyang, Henan
  - Nanyang Second General Hospital, Nanyang, Henan
  - First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - The Third People's Hospital of Hubei Province, Wuhan, Hubei
  - Hunan Provincial People's Hospital, Changsha, Hunan
  - Sinapharm North Hospital, Baotou, Inner Mongolia
  - Ordos Central Hospital, Ordos, Inner Mongolia
  - Tongliao City Hosptial, Tongliao, Inner Mongolia
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Jiangxi Provincial People's Hospital, Nanchang, Jiangxi
  - Shandong Provincial Hospital, Jinan, Shandong
  - Shandong Provincial Qianfoshan Hospital, Jinan, Shandong
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Beichen Hospital of Traditional Chinese Medicine, Tianjin, Tianjin Municipality
  - TEDA Hospital, Tianjin, Tianjin Municipality

REFERENCES:
- [Background] Wu C, Sun C, Wang L, Lian Y, Xie N, Huang S, Zhao W, Ren M, Wu D, Ding J, Song H, Wang Y, Ma Q, Ji X. Low-Dose Tirofiban Treatment Improves Neurological Deterioration Outcome After Intravenous Thrombolysis. Stroke. 2019 Dec;50(12):3481-3487. doi: 10.1161/STROKEAHA.119.026240. Epub 2019 Oct 1. PMID 31570084
- [Result] Zhao W, Che R, Shang S, Wu C, Li C, Wu L, Chen J, Duan J, Song H, Zhang H, Ling F, Wang Y, Liebeskind D, Feng W, Ji X. Low-Dose Tirofiban Improves Functional Outcome in Acute Ischemic Stroke Patients Treated With Endovascular Thrombectomy. Stroke. 2017 Dec;48(12):3289-3294. doi: 10.1161/STROKEAHA.117.019193. Epub 2017 Nov 10. PMID 29127270
- [Derived] Wang J, Qiao Y, Li S, Li C, Wu C, Wang P, Yang T, Ji X, Ma Q, Zhao W. Effects of tirofiban in preventing neurological deterioration in acute ischemic stroke with intracranial artery stenosis: A post hoc analysis of the TREND Trial. Eur Stroke J. 2025 Sep;10(3):919-928. doi: 10.1177/23969873251319151. Epub 2025 Feb 14. PMID 39950764
- [Derived] Wang J, Li S, Li C, Wu C, Song H, Ma Q, Ji X, Zhao W; TREND Investigators. Safety and efficacy of tirofiban in preventing neurological deterioration in acute ischemic stroke (TREND): Protocol for an investigator-initiated, multicenter, prospective, randomized, open-label, masked endpoint trial. Brain Circ. 2024 Jun 26;10(2):168-173. doi: 10.4103/bc.bc_93_23. eCollection 2024 Apr-Jun. PMID 39036300
- [Derived] Zhao W, Li S, Li C, Wu C, Wang J, Xing L, Wan Y, Qin J, Xu Y, Wang R, Wen C, Wang A, Liu L, Wang J, Song H, Feng W, Ma Q, Ji X; TREND Investigators. Effects of Tirofiban on Neurological Deterioration in Patients With Acute Ischemic Stroke: A Randomized Clinical Trial. JAMA Neurol. 2024 Jun 1;81(6):594-602. doi: 10.1001/jamaneurol.2024.0868. PMID 38648030